CLINICAL TRIAL: NCT00227630
Title: A Phase II Feasibility Trial of Induction Chemotherapy Followed by Extrapleural Pneumonectomy and Postoperative Radiotherapy in Patients With Malignant Pleural Mesothelioma
Brief Title: Pemetrexed Disodium and Cisplatin Followed By Surgery and Radiation Therapy in Treating Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: EORTC-08031; EORTC-08031; 2004-004273-28 (EudraCT Number)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Malignant Mesothelioma
Keywords: epithelial mesothelioma; sarcomatous mesothelioma; localized malignant mesothelioma; recurrent malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Cisplatin; Pemetrexed; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: pemetrexed disodium
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pemetrexed disodium and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pemetrexed disodium may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy before surgery may shrink the tumor so that it can be removed. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving pemetrexed disodium and cisplatin followed by surgery and radiation therapy works in treating patients with malignant pleural mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of neoadjuvant chemotherapy comprising pemetrexed disodium and cisplatin followed by extrapleural pneumonectomy and high-dose postoperative 3D-conformal radiotherapy, in terms of 90-day progression-free survival, in patients with malignant pleural mesothelioma.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine progression-free survival and overall survival of patients treated with this regimen.

OUTLINE: This is a non-randomized, multicenter study.

* Neoadjuvant chemotherapy: Patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 2 hours on day 1. Treatment repeats every 3 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients are evaluated 3 weeks after completion of neoadjuvant chemotherapy. Patients without disease progression proceed to surgery.
* Extrapleural pneumonectomy: Within 21-56 days after completion of neoadjuvant chemotherapy, patients undergo extrapleural pneumonectomy. Patients are evaluated 30 days after surgery. Patients without disease progression undergo high-dose 3D-conformal radiotherapy.
* High-dose 3D-conformal radiotherapy: Beginning 30-84 days after surgery, patients undergo high-dose 3D-conformal radiotherapy daily for 30 days.

After completion of study treatment, patients are followed on days 42 and 90, every 3 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 52 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant pleural mesothelioma

  * All subtypes allowed
* T1-3, N0-1, M0 disease

  * No N2 or N3 involvement confirmed by mediastinoscopy within 21 days before study entry
* No clinical invasion of mediastinal structures (e.g., heart, aorta, spine, esophagus)
* No wide-spread chest wall invasion except focal chest wall lesions
* No clinical or radiological evidence of shrinking hemithorax
* No clinically significant third-space fluid (e.g., pleural effusions or ascites) that cannot be managed with thoracentesis or pleurodesis

PATIENT CHARACTERISTICS:

Age

* Under 70

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC > 3,500/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin ≥ 11 g/dL

Hepatic

* AST and ALT < 1.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Alkaline phosphatase < 1.5 times ULN

Renal

* Creatinine clearance ≥ 60 mL/min
* Acceptable (predicted) post-radiotherapy renal function by semiquantitative isotope renography, with a relative contribution of the contralateral kidney of ≥ 40%

Pulmonary

* See Disease Characteristics

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Deemed to be fit enough to undergo study treatment
* No preexisting sensory neurotoxicity > grade 1
* No uncontrolled infection
* No prior or concurrent melanoma, breast cancer, or hypernephroma
* No other malignancy within the past 5 years except carcinoma in situ of the cervix or adequately treated basal cell skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy
* No concurrent routine use of colony-stimulating factors during neoadjuvant chemotherapy

  * Concurrent secondary prophylactic use allowed during neoadjuvant chemotherapy
* No concurrent secondary prophylactic use of colony-stimulating factors during post-operative radiotherapy

Chemotherapy

* No prior chemotherapy for mesothelioma

Endocrine therapy

* No concurrent hormonal cancer therapy

Radiotherapy

* No prior radiotherapy to the lower neck, thorax, or upper abdomen

Surgery

* See Disease Characteristics

Other

* No other concurrent anticancer therapy
* No other concurrent experimental medications
* No nonsteroidal anti-inflammatory drugs or salicylates for 2 days before, during, and 2 days after administration of neoadjuvant chemotherapy (5 days before and 2 days after for drugs with a long half-life [e.g., naproxen, piroxicam, diflunisal, or nabumetone])

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2005-07; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Feasibility in terms of 90-day progression-free survival

SECONDARY OUTCOMES:
Toxicity
Progression-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Paul Van Schil, MD, PhD, Study Chair — University Hospital, Antwerp
Locations (8):
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- Italy (3):
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Azienda Ospedaliera Di Parma, Parma
  - Universita Degli Studi di Udine, Udine
- Netherlands (2):
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
- United Kingdom (2):
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland

REFERENCES:
- [Result] O'Brien ME, Konopa K, Lorigan P, Bosquee L, Marshall E, Bustin F, Margerit S, Fink C, Stigt JA, Dingemans AM, Hasan B, Van Meerbeeck J, Baas P. Randomised phase II study of amrubicin as single agent or in combination with cisplatin versus cisplatin etoposide as first-line treatment in patients with extensive stage small cell lung cancer - EORTC 08062. Eur J Cancer. 2011 Oct;47(15):2322-30. doi: 10.1016/j.ejca.2011.05.020. Epub 2011 Jun 16. PMID 21684151
- [Result] Van Schil PE, Baas P, Gaafar R, Maat AP, Van de Pol M, Hasan B, Klomp HM, Abdelrahman AM, Welch J, van Meerbeeck JP; European Organisation for Research and Treatment of Cancer (EORTC) Lung Cancer Group. Trimodality therapy for malignant pleural mesothelioma: results from an EORTC phase II multicentre trial. Eur Respir J. 2010 Dec;36(6):1362-9. doi: 10.1183/09031936.00039510. Epub 2010 Jun 4. PMID 20525721